CLINICAL TRIAL: NCT01920139
Title: Ultrasound Guided Core Biopsy vs Fine Needle Aspiration for Evaluation of Axillary Lymphadenopathy in Patients Suspected of Having Breast Cancer.
Brief Title: Ultrasound Guided Core Biopsy vs Fine Needle Aspiration for Evaluation of Axillary Lymphadenopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Suros Surgical (now Hologic ) (Unknown)
Responsible Party: Principal Investigator, Marie Ganott, MD, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PRO07100450
Record Dates: First submitted 2013-08-01; First posted 2013-08-09 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-08

CONDITIONS: Focus: Breast Cancer With Axillary Node Metastasis
MeSH Terms: interventions — Biopsy, Fine-Needle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Breast cancer and Axillary Adenopathy (Other): Women with breast cancer with abnormal appearing ipsilateral axillary nodes undergoing fine needle aspiration and core biopsy of a lymph node.
  Interventions: Procedure: Fine needle aspiration and core biopsy of lymph node; Procedure: Axillary surgery; Other: Titanium marker

INTERVENTIONS:
Procedure: Fine needle aspiration and core biopsy of lymph node — Ultrasound guided fine needle aspiration of an abnormal lymph node followed by ultrasound guided core biopsy of the same node followed by clip placement into the node.
Procedure: Axillary surgery — Patients underwent axillary node dissection or excision of setinel axillary nodes at the time of surgical treatment of their breast cancer.
Other: Titanium marker — A titanium marker was deposited into the lymph node that was percutaneously biopsied , immediately after the last tissue sample obtained.

SUMMARY:
The study was performed to determine if either ultrasound guided core biopsy or fine needle aspiration of an axillary lymph node has superior sensitivity in detecting metastatic carcinoma from the ipsilateral breast.

DETAILED DESCRIPTION:
Women with suspected or recently diagnosed breast cancer and ipsilateral abnormal appearing axillary lymph nodes underwent fine needle aspiration immediately followed by core biopsy of the same lymph node.Cytology results from the fine needle aspiration (FNA)and histology from the core biopsy were compared to surgical pathology from axillary node excision to determine if either method of percutaneous node sampling was more sensitive in detecting metastasis. Pain during each procedure was also compared.

ELIGIBILITY:
Inclusion Criteria:

* Women with breast cancer and abnormal ipsilateral axillary nodes visible on sonography.

Exclusion Criteria:

* Inability to understand consent form.
* Emotionally unprepared to discuss possibility of axillary metastasis
* Node not amenable to core biopsy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2008-12; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Fraction of metastatic nodes found at axillary surgery that were identified pre-surgically by FNA vs. core biopsy | 1 week to 10 months
  Results of FNA cytology and core biopsy histology are compared to axillary surgery results.

OTHER OUTCOMES:
Pain associated with each type of percutaneous biopsy procedure | immediate at time of biopsy
  Patients were asked to report pain level during the 2 types of percutaneous biopsy.

CONTACTS AND LOCATIONS:
Locations (1):
- Magee Womens Hospital, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Ganott MA, Zuley ML, Abrams GS, Lu AH, Kelly AE, Sumkin JH, Chivukula M, Carter G, Austin RM, Bandos AI. Ultrasound Guided Core Biopsy versus Fine Needle Aspiration for Evaluation of Axillary Lymphadenopathy in Patients with Breast Cancer. ISRN Oncol. 2014 Feb 4;2014:703160. doi: 10.1155/2014/703160. eCollection 2014. PMID 24649373